CLINICAL TRIAL: NCT00961688
Title: The Impact of PCOS on Quality of Life and Healthcare Beliefs
Brief Title: The Impact of Polycystic Ovary Syndrome (PCOS) on Quality of Life and Healthcare Beliefs
Acronym: PCOS
Status: Completed | Type: Observational
Sponsor: Georgia Reproductive Specialists (Other)
Responsible Party: Mark Perloe, M.D., Georgia Reproductive Specialists
Other Study IDs: GRS-3296
Record Dates: First submitted 2009-08-14; First posted 2009-08-19 (Estimated); Last update posted 2010-02-03 (Estimated); Status verified 2010-02

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS; polycystic ovary syndrome; Polycystic ovarian syndrome; infertility; ovulation
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
Women with Polycystic Ovary Syndrome (PCOS) between the age of 18 and 55 are being recruited to participate in an online survey to determine the impact of PCOS on quality of life and interaction with the healthcare system. This online survey will take 15-20 minutes to complete. Participants will receive no direct benefit, but the information provided will contribute to the knowledge of this condition and the development of improved healthcare for women with PCOS. For more information or to participate in this study, please visit http://pcossurvey.vze.com

ELIGIBILITY:
Inclusion Criteria:

* Women with Polycystic Ovary Syndrome (PCOS) between the age of 18 and 55

Exclusion Criteria:

* N/A

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with Polycystic Ovary Syndrome (PCOS) between the age of 18 and 55
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Perloe, MD, Principal Investigator — Georgia Reproductive Specialists
Locations (1):
- Georgia Reproductive Specialists, Atlanta, Georgia, United States

REFERENCES:
- See also: Link to online PCOS Survey — http://pcossurvey.vze.com